CLINICAL TRIAL: NCT00464997
Title: The Effect of Low Dose Aspirin on the Pharmacokinetics of Methotrexate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: TASMC-07-OE-156-CTIL
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Rheumatoid Arthritis
Keywords: methotrexate aspirin pharmacokinetics
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
High dose aspirin have been shown to increase the level of Methotrexat in patients with Rheumatoid Arthritis. However, most of RA patients are not currently treated with high dose aspirin. On the other hand, they frequently receive treatment with low dose aspirin. The effect of low dose aspirin on the levels of Methotrexate is not well known. Therefore,the purpose of this study is to assess the effect of low dose aspirin on the levels of methotrexate.

DETAILED DESCRIPTION:
Thirty Rheumatoid Arthritis patients currently treated with low dose methotrexate (MTX) will participate in this study. On the day of intake of methotrexate, the patients will receive 10 mg of MTX. Serum levels of MTX will be measured at time 0,30 ,90, 120 minutes, and after 12 and 24 hours.

Two weeks later, the patients will be recommended to take 100 mg aspirin/d during a week. The levels of MTX will be measured after a week of treatment in a way similar to a week before.

ELIGIBILITY:
Inclusion Criteria:

* RApatients treated with Methotrexate

Exclusion Criteria:

* Contraindication to aspirin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2007-06

CONTACTS AND LOCATIONS:
Overall Officials: Ori Elkayam, M.D, Principal Investigator — Tel Aviv Medical Center